CLINICAL TRIAL: NCT01613820
Title: Combination of Anticholinergic and Glutamatergic Effects in Treatment-resistant Major Depressive Disorder. A Pilot Study
Brief Title: Ketamine and Scopolamine Infusions for Treatment-resistant Major Depressive Disorder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Cristina Cusin, MD, Instructor HMS, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-P-000624
Record Dates: First submitted 2012-05-31; First posted 2012-06-07 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Ketamine; Scopolamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ketamine plus placebo (Experimental): Subjects assigned to this paradigm will receive a 15 minute infusion of normal saline (placebo) followed by IV ketamine at 0.25mg/kg over 45 minutes twice a week for 3 weeks.
  Interventions: Drug: Ketamine
- Scopolamine plus placebo (Experimental): Subjects will receive a 15 minute infusion of IV scopolamine 2ug/kg followed by a 45 minute infusion of normal saline (placebo).
  Interventions: Drug: Scopolamine
- Ketamine plus scopolamine (Experimental): Subject will receive an IV scopolamine infusion at a dose of 2ug/kg over 15 minutes, followed by an IV infusion of ketamine at a dose of 0.25mg/kg over 45 minutes.
  Interventions: Drug: Ketamine; Drug: Scopolamine

INTERVENTIONS:
Drug: Ketamine — ketamine IV 0.25mg/kg infusions twice a week for 3 weeks as augmentation of ongoing antidepressant regimen.
  Arms: Ketamine plus placebo; Ketamine plus scopolamine
Drug: Scopolamine — Scopolamine 2ug/kg over 15 minutes twice a week for 3 weeks as augmentation of ongoing antidepressant regimen
  Arms: Ketamine plus scopolamine; Scopolamine plus placebo

SUMMARY:
Ketamine infusions resulted in an acute reduction in global depression scores and in severity of suicidal ideation. Scopolamine infusions produced also a significant improvement in depression that was sustained over time.

We therefore plan to investigate the feasibility and efficacy of open-label repeated intravenous administration of ketamine and scopolamine combined in this population of severely depressed, treatment-resistant patients. The results from this study could lead to the development of new strategies for the treatment of patients with TRD.

DETAILED DESCRIPTION:
Patients will undergo two weeks of prospective observation, they will then receive IV infusions of ketamine, scopolamine or both per randomization as augmentation of their ongoing antidepressant regime. The schedule of administration will be twice a week of three weeks. After this phase the subject will be followed with assessments every two weeks for three months.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with sever treatment-resistant depression
* Currently depressed
* Currently under regular psychiatric care
* On an aggressive antidepressant regimen, stable for 4 weeks

Exclusion Criteria:

* No history of other major psychiatric illnesses, including bipolar disorder
* No history of psychosis
* No history of drug abuse
* No major medical illness or unstable medical condition.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale - 28 items | up to 4 months
  Subjects will be assessed with HAMD-28

SECONDARY OUTCOMES:
Systematic Assessment for Treatment Emergent Events (SAFTEE) | up to 4 months
  Subjects will be monitored for emergence of side effects weekly for the first 8 weeks, then every two weeks for 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Cusin, M.D., Principal Investigator — MGH Department of Psychiatry
Locations (1):
- Depression Clinical and Reseach Program - MGH, Boston, Massachusetts, United States